CLINICAL TRIAL: NCT03389932
Title: Working Within an Integrated Learning Healthcare System to Improve Living Kidney Donation Knowledge Across the CKD Continuum for All Racial Groups
Brief Title: Explore Transplant @Home Within Kaiser Permanente Southern California
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Amy D. Waterman, Director, Patient Engagement, Diversity, and Education, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R39OT29879
Record Dates: First submitted 2017-12-26; First posted 2018-01-04 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Control) (No Intervention): For patients who are randomized to the control condition and who are or become potentially eligible for transplant during their enrollment in the study, they will not receive any additional interventions during the study period. Patients in this condition will only receive the education that is administered by the KPSC Kidney Transplant Program and will not receive any educational materials designed for the intervention group of this study.
- Patient-Guided (Experimental): Patients in the ET@Home study condition will receive four modules of video and print transplant education over a 6-month period. After each module is mailed, 3 postcards are mailed weekly that recap important transplant educational content covered within the videos. Patients will have the opportunity to participate in a texting component of ET@Home that also sends small pieces of educational content and learning reminders by phone each week.
  Interventions: Behavioral: Patient-Guided

INTERVENTIONS:
Behavioral: Patient-Guided — Patients in the ET@Home study condition will receive four modules of video and print transplant education over a 6-month period. After each module is mailed, 3 postcards are mailed weekly that recap important transplant educational content covered within the videos. Patients will have the opportunity to participate in a texting component of ET@Home that also sends small pieces of educational content and learning reminders by phone each week.
  Arms: Patient-Guided

SUMMARY:
Today, there are 25 million Americans with chronic kidney disease (CKD) and 660,000 patients in full kidney failure, the final CKD stage, known as end stage renal disease (ESRD). Over half of ESRD patients are Black, Hispanic, or Asian. ESRD patients must either receive regular dialysis treatments, by which waste is filtered from the blood by a machine, or a kidney transplant from a deceased or living donor. Five-year survival on dialysis is only 40%, compared to 74% with a deceased donor kidney transplant (DDKT) and 87% with a living donor kidney transplant (LDKT). Despite the known health benefits of DDKT and LDKT, 70% of ESRD patients remain on dialysis, especially ethnic/racial minorities.

An American Society of Transplantation (AST) Consensus Conference recently recommended that patients in all CKD stages should have the opportunity to learn about and decide which treatment option is right for them, particularly about LDKT. However, early education about LDKT and DDKT is inconsistent and often poor, with early stage CKD patients and ethnic/racial minorities even less likely to receive it.

Through previous HRSA grants, Dr. Waterman designed the Explore Transplant@Home (ET@Home) video-guided education program, and found that it significantly increased LDKT knowledge and informed decision-making for Black and White dialysis patients in Missouri when delivered by mail and supported through bimonthly postcards and texting. Now based at the University of California, Los Angeles (UCLA), she has partnered with Kaiser Permanente Southern California (KPSC), an integrated learning healthcare system providing insurance coverage and comprehensive care to 65,000 patients in CKD Stages 3, 4 and 5 (ESRD) (24% Hispanic, 52% White, 15% Black, and 9% Asian; 10% Spanish-speaking).

DETAILED DESCRIPTION:
Today, there are 25 million Americans with chronic kidney disease (CKD) who are at risk for kidney failure and 660,000 patients with end-stage renal disease (ESRD). To sustain life, ESRD patients, among whom 31% are Black, 15% are Hispanic, and 5% are Asian, must either receive daily or weekly dialysis treatments, by which waste is filtered from the blood by a machine, or receive a kidney transplant from a deceased or living donor. Five-year survival for patients on dialysis is only 40%, compared to 74% for patients who receive a deceased donor kidney transplant (DDKT) and 87% for patients who receive a living donor kidney transplant (LDKT)1. Patients who receive kidney transplants live 5-15 years longer than if they remained on dialysis, and have a better health-related quality of life (HRQOL), including a greater likelihood of being in the workforce during their critical earning years2. While LDKT is the medically optimal and most cost effective renal replacement therapy (RRT) for patients with ESRD, LDKT rates have declined by 17% from 2004-2014. In 2014, in the U.S., 17,106 patients received a transplant (5,536 LDKTs) while 8,021 patients also died or became too ill to remain on the list, 70% of whom were racial/ethnic minorities. Of the 2,039 transplants performed in California in 2014, only 595 were from living donors (OPTN data as of 12/11/2015).

Since kidneys often fail slowly over months or years, a patient's level of kidney function is monitored over time as it decreases in nephrologists' offices nationwide. As recommended by a recent American Society of Transplantation (AST) Consensus Conference, all patients in Stage 3 (Moderate CKD), Stage 4 (Severe CKD), or Stage 5 (End Stage CKD) should receive comprehensive education about DDKT and LDKT, especially racial/ethnic minorities. Once patients reach ESRD and begin dialysis, established CKD and Centers for Medicare and Medicaid Services (CMS) guidelines recommend that dialysis patients be educated about their RRT options, the medical risks involved, and the advantages to transplant so that they can make informed RRT decisions4. Since transplants received within the first 6 months of beginning dialysis result in the best health outcomes,5 one Healthy People 2020 goal is to, "Increase the proportion of dialysis patients wait-listed and/or receiving a deceased donor kidney transplant within one year of ESRD start (among patients under 70 years of age)." Unfortunately, research has shown that many patients in CKD clinics are inconsistently educated about LDKT, particularly patients who are socioeconomically disadvantaged or members of racial/ethnic minority groups.

Without a nationally-coordinated healthcare system, it is extremely difficult to ensure that kidney patients in Stages 3-5 who are served by different health practitioners and organizations all learn about DDKT and LDKT and make informed treatment decisions. Providers also report having limited time to educate about transplant outside of transplant centers and inadequate educational materials. Thus, disseminating transplant education within a large health care system, with its fully integrated care management program, diverse membership, and ability to track a large patient population across the entire course of their kidney disease, may be an opportune way to educate large numbers of diverse patients about the opportunities for and risks and benefits of living kidney donation.

Kaiser Permanente Southern California (KPSC) is a large, integrated healthcare system providing coverage and care to over 4 million members throughout Los Angeles, San Diego,Kern, San Bernardino, Riverside, and Ventura Counties. KPSC provides coverage to nearly 65,000 patients with CKD stages 3-5. About 24% of these patients are Hispanic, 52% White, 15% Black, and 9% Asian, similar to the broader CKD population in California.

First, this team will conduct extensive qualitative and quantitative formative research to understand and compare the knowledge, informed decisionmaking and educational needs of these diverse patient groups prior to intervention. Second, they will design a Spanish-language version of ET@Home. Third, they will conduct a randomized controlled trial (RCT) of 1,200 Black, Hispanic, Asian, and White patients in CKD Stages 3-5 where patients will be randomized to receive: (1) no additional education other than what is provided within KPSC (standard-of-care); or (2) a video-guided, four-part ET@Home program delivered by mail and supported through bimonthly postcards and texting over six months. The study aims and hypotheses are as follows: Aim 1: Using qualitative methodology, to assess the LDKT educational needs of CKD Stage 3-5 patients and their support networks by race/ethnicity and primary language spoken.

Hypothesis 1: CKD Stage 3-5 patients and their support networks will have varying needs for educational content about LDKT based on their race/ethnicity and primary language spoken.

Hypothesis 2: Providers will identify important patient needs for LDKT educational content and opportunities for improvement within the KPSC transplant educational system.

Aim 2: Before intervention, to assess differences in knowledge and decision-making about the opportunities for and risks and benefits of living kidney donation for 1200 CKD Stage 3-5 patients by race/ethnicity and primary language spoken.

Hypothesis: Patients earlier in the CKD continuum, patients who speak Spanish, and non- White patients will have less knowledge about the opportunities for and risks and benefits of living kidney donation and will be making less informed LDKT decisions.

Aim 3: Compared to KPSC education, to conduct a randomized controlled trial in English and Spanish of ET@Home for CKD Stage 3-5 patients to assess its effectiveness to increase LDKT knowledge and decision-making by race/ethnicity and primary language spoken.

Hypothesis 1: At the conclusion of the trial, CKD patients who receive ET@Home will have greater transplant knowledge and be more likely to make an informed treatment decision than patients receiving KPSC education alone.

Hypothesis 2: ET@Home will be more or equally effective for patients earlier in the CKD continuum, patients who speak Spanish, and non-White patients than patients in these subgroups receiving KPSC education alone.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be at least 18 years of age.
2. Participant must self-identify as African American, White, Hispanic, or Asian.
3. Participant must currently be classified as having CKD 3, 4 or 5.
4. Participant must be able to speak and read in English or Spanish.

Exclusion Criteria:

1. Participant is not classified as having CKD 3,4, or 5.
2. Participant cannot speak or read in English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 977 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Deceased Donor Kidney Transplant (DDKT) and Living Donor Kidney Transplant (DDKT) Knowledge | 6 months
  Patients will be asked true/false and multiple choice questions to determine their level of knowledge regarding basic facts, advantages, risks and outcomes of DDKT and LDKT (e.g., "Patients older than 75 years can receive transplants"; "Compared to transplants from donors who have died, how long do transplants from living donors last?"). Scores for this scale are created by summing the number of correct answers given by the patient, creating a theoretical range of 0-25 with higher scores indicating more knowledge.

SECONDARY OUTCOMES:
Decisional Balance | 6 months
  Decisional Balance will be measured for DDKT (DB-DDKT) and for LDKT (DB-LDKT). DB-DDKT, a measure of a patient's perception of the benefits and disadvantages of deceased donor kidney transplant. This measure has been validated in a sample of dialysis patients84. Both measures contain two subscales, Pros and Cons of 6 items, wherein patients rate the importance of a specific Pro or Con to their DDKT or LDKT decision-making (e.g., "I would not have to be on dialysis") on a Likert-type scale from (1) "Not important" to (5) "Extremely important". Scores for the subscales will be obtained by summing the patients' responses to the items, implying a theoretical range of 6-30, with higher scores indicating more Pros or Cons, depending on the subscale. The DB-LDKT was also recently validated in a sample of dialysis patients.
Informed Decision-Making | 6 months
  Informed Decision-Making will be assessed in two ways. First, patients will be asked the following three questions: "I have all the facts I need to make an informed decision about whether to pursue DDKT/LKDT/remain on dialysis" (agree/disagree). Each of these questions will be treated as individual items and analyzed separately as outcomes.
  We will also use a validated measure of decisional conflict, the Decisional Conflict Scale (DCS). This scale assesses factors contributing to patients' uncertainty in making health-related decisions, and patients' assessment of their perceived effective decision-making. Each of these dimensions of decisional conflict will be considered as subscales, and together they will be considered as a total decisional conflict measure. The entire scale has 16 items (3 for decision uncertainty, 9 for factors contributing to uncertainty, and 4 for effective decision-making), each measured on a scale of (1) strongly agree to (5) strongly disagree.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Research and Evaluation, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waterman AD, Anderson C, Alem A, Peipert JD, Beaumont JL, Henry SL, Dub B, Ambriz L, Bijjala N, Lipsey AF, Mittman B. A randomized controlled trial of Explore Transplant at Home to improve transplant knowledge and decision-making for CKD 3-5 patients at Kaiser Permanente Southern California. BMC Nephrol. 2019 Mar 4;20(1):78. doi: 10.1186/s12882-019-1262-9. PMID 30832619